CLINICAL TRIAL: NCT04736277
Title: The Effect of HbA1c on Perioperative Neurocognitive Disorders in Patients Undergoing Elective Non-cardiac Surgery Under General Anesthesia.
Brief Title: HbA1c and Neurocognitive Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Collaborators: University Hospital, Ioannina (Other); Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: HbA1c and NCD
Record Dates: First submitted 2020-10-24; First posted 2021-02-03 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-04

CONDITIONS: Neurocognitive Disorders; HbA1c
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Noncardiac surgery: Documentation of HbA1c in patients undergoing noncardiac surgery under general anesthesia
  Interventions: Other: Preoperative HbA1c

INTERVENTIONS:
Other: Preoperative HbA1c — Documentation of the preopetative HbA1c in patients undergoing noncardiac surgery under general anesthesia

SUMMARY:
Preliminary evidence suggest a possible relationship between HbA1c and perioperative neurocognitive disorders (NCD). We are going to investigate whether the preoperative value of HbA1c in patients undergoing elective non-cardiac surgery under general anesthesia, are related with increased risk of perioperative NCD.

DETAILED DESCRIPTION:
It is estimated that approximately 10% of elderly undergoing surgery will develop cognitive changes perioperatively, while in some reports the incidence rises up to 80%. Despite the reported high prevalence of perioperative neurocognitive disorders (NCD), their exact etiology is still largely unknown.

Preliminary evidence suggest a possible relationship between HbA1c and perioperative neurocognitive disorders (NCD). We are going to investigate whether the preoperative value of HbA1c in patients undergoing elective non-cardiac surgery under general anesthesia, are related with increased risk of perioperative NCD.

ELIGIBILITY:
Inclusion Criteria:

* 1) 45 - 80 years
* 2) American Society of Anesthesiologists physical status I to III
* 3) elective general, urological, gynecological and orthopedic surgery under general anesthesia
* 4) native speakers of the Greek language

Exclusion Criteria:

* 1) refused to participate or sign the informed consent form
* 2) had undergone surgery or anesthesia within the last 30 days
* 3) had any prior or current history involving an affliction of the central nervous system
* 4) were diagnosed with severe cognitive decline based on the 16 - item Informant Questionnaire on Cognitive Decline (IQCODE - 16)
* 5) suffered from severe hearing or visual impairment
* 6) any psychiatric disorder
* 7) had a score >5 in the Geriatric Depression Scale (GDS - 15)
* 8) or a score in females < 4 males < 2 in the Lawton - Brody Instrumental Activities of Daily Living Scale (I.A.D.L.)
* 9) reported alcohol consumption > 35 units/week
* 10) drug dependence
* 11) had undergone previous neuropsychological testing
* 12) Diabetes Mellitus type II with > 10 years of diagnosis
* 13) Diabetes Mellitus type I
* 14) Hemoglobin A1c (HbA1c) > 7.5%
* 15) suffered from hemodynamical instability (> 20% alterations of blood pressure perioperatively)
* 16) or desaturation (one or more events of SpO2 < 80% for more than 2 minutes) peri-operatively
* 17) or blood loss of more than one unit

Ages: 45 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - All patients 45 - 80 years old, ASA I-III undergoing elective general, urological, gynecological and orthopedic surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Neurocognitive Disorders assessed with CAM | 1st postoperative day
  Screening for POD assessed with CAM
Incidence of Postoperative Neurocognitive Disorders with IQCODE-16 | 10th postoperative day
  Screening for POCD with IQCODE-16
Incidence of Postoperative Neurocognitive Disorders with IQCODE-16 | 3 months postoperatively
  Screening for POCD with IQCODE-16
Incidence of Postoperative Neurocognitive Disorders with IQCODE-16 | 6 months postoperatively
  Screening for POCD with IQCODE-16
Incidence of Postoperative Neurocognitive Disorders with IQCODE-16 | 9 months postoperatively
  Screening for POCD with IQCODE-16

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, MD, PhD, Study Chair — Professor of Anesthesiology; Maria Ntalouka, MD, PhD, Principal Investigator — Consultant of Anesthesiology
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided